CLINICAL TRIAL: NCT01254903
Title: Phase I Study of Feasibility of Single Session Spine Stereotactic Radiosurgery (SSRS) in the Primary Management in Patients With Inoperable, Previously Unirradiated Metastatic Epidural Spinal Cord Compression (MESCC)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0655; NCI-2011-00269 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-12-03; First posted 2010-12-07 (Estimated); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Epidural Spinal Cord Compression
Keywords: Stereotactic Radiosurgery; Radiation; Radiotherapy; Metastatic Epidural Spinal Cord Compression; MESCC
MeSH Terms: interventions — Radiosurgery; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stereotactic Radiosurgery (SSRS) (Experimental): Target dose of 18 or 24 Gy to spine in single session of radiation treatment.
  Interventions: Procedure: Stereotactic Radiosurgery (SSRS)

INTERVENTIONS:
Procedure: Stereotactic Radiosurgery (SSRS) — Target dose of 18 or 24 Gy to spine in single session of radiation treatment.
  Other Names: Radiotherapy; Radiation therapy

SUMMARY:
The goal of this clinical study is to learn the feasibility of using a single session of radiation, known as spine stereotactic radiosurgery (SSRS), to treat metastatic epidural spinal cord compression.

DETAILED DESCRIPTION:
Spinal cord compression is often treated with surgery followed by radiation in small doses everyday for a number of days. When a patient cannot or will not have surgery, radiation is given daily. With increased accuracy and precision, higher doses of radiation can be given in a single session. Giving a higher dose in a single session may increase the chance that the tumor will stop growing into the spinal canal and will prevent spinal cord injury. This study will also help to identify the tolerance of the spinal cord to radiation in a single session.

Spine Stereotactic Radiosurgery:

You will lie in the mold that was made for you for 45-120 minutes while you receive your radiation treatment.

Follow-up Visits:

You will have follow-up visits at Months 3 (+/-2 weeks ), 6 (+/-4 weeks), 9 (+/-4 weeks), 12 (+/-8 weeks), 18 (+/-8 weeks), and 24 (+/-8 weeks) and then every 6 months after that. At each follow-up visit:

* Your medical history will be recorded, including any use of steroids.
* You will have a neurological exam.
* You will complete the 3 questionnaires about health, symptoms you may be having, and about pain.
* You will have an MRI of the spine (except for Month 1).

If you are unable to return for follow-up clinic visits, you will be called and asked about your medical history, and you will complete the 3 questionnaires about your health, symptoms you may be having, and about pain. This call should take about 20 minutes.

Length of Study:

Your treatment will last 1 day. You will continue having follow-up visits or phone calls for as long as possible.

This is an investigational study. SSRS is FDA approved. The use of SSRS to treat metastatic epidural spinal cord compression is investigational.

Up to 36 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Greater than or equal to 18 years old
2. Radiographically documented metastatic epidural compression on spine Magnetic resonance imaging (MRI) within 4 weeks of registration, defined radiographically, ranging from minimal canal compromise and thecal indentation to actual displacement of the spinal cord.
3. Maximum of 3 contiguous vertebral levels involved with metastasis in the spine to be irradiated in a single session
4. Signed Informed consent
5. Diagnosis of cancer (not one of the more radiosensitive histologies, see exclusion criteria) including but not limited to non-small cell lung cancer, breast, prostate, renal cell, melanoma, gastrointestinal, sarcoma, thyroid, head and neck primary, and unknown primary tumors
6. Motor Strength >/= 4 out of 5 in extremity or extremities affected by the level of the spinal cord compression
7. Karnofsky performance status (KPS) >/= 40
8. Patients deemed to be inoperable by patient refusal, by neurosurgical evaluation, or for any reason

Exclusion Criteria:

1. Patient with radiosensitive histologies (lymphoma, multiple myeloma, small cell carcinoma, germ cell tumors) as conventional radiation is likely to be effective
2. Prior irradiation of the spine site and level to be treated
3. Inability to tolerate lying flat on treatment table for greater than 30 minutes.
4. Patients unable to undergo MRI of the spine
5. Patients who are pregnant
6. Patients who have cord compression from bone components or configuration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2010-12-03 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of Occurrences of Paralysis caused by Radiation Myelitis (RM) | Up to 12 months following radiation
  Incidence of patients who are ambulatory at baseline, 3 months and 6 months will be tabulated. Cases of patients who develop spinal cord myelopathy determined to be radiation related graded according to NCI CTC v4.0 scale.

CONTACTS AND LOCATIONS:
Overall Officials: Amol J. Ghia, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org